CLINICAL TRIAL: NCT01380197
Title: Choosing Opioid Management for Pain and Analyzing ACS Rates Equally
Brief Title: Choosing Opioid Management for Pain and Analyzing Acute Chest Syndrome (ACS) Rates Equally
Acronym: COMPARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Healthcare of Atlanta (Other)
Collaborators: Atlanta Clinical and Translational Science Institute (Other)
Responsible Party: Principal Investigator, Saadia Khizer, Iris Buchanan MD, Children's Healthcare of Atlanta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-076
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-01

CONDITIONS: Pain; Sickle Cell Disease
Keywords: pain; sickle cell; nubain; morphine; acute chest; side effects
MeSH Terms: conditions — Pain; Anemia, Sickle Cell | interventions — Morphine; Nalbuphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Randomizing particiipants to Morphine (Active Comparator): Randomizing participants to Morphine or Nubain for treatment of Sickle Cell Pain Crisis
  Interventions: Drug: Morphine
- Randomization to Nubain (Active Comparator): Randomization toNubain or Morphine for the management of Pain Crisis in Sickle Cell patients
  Interventions: Drug: Nubain

INTERVENTIONS:
Drug: Morphine — Loading Dose: 0.1mg/kg. May repeat every 15 min up to a maximum of 3 total doses until pain controlled.
  Continuous rate: 0.01-0.04mg/kg/hr (titrated to comfort level) PCA dose 0.01-0.03 mg/kg maximum 1.6 mg/dose 4 hour dose limit 0.24-0.3 mg/kg (Maximum dosing will not exceed 25 mg/4 hrs).
  Arms: Randomizing particiipants to Morphine
Drug: Nubain — Loading Dose: 0.1mg/kg. May repeat every 15 min up to a maximum of 3 total doses until pain controlled.
  Continuous rate: 0.01-0.04mg/kg/hr (titrated to comfort level) PCA dose 0.01-0.03 mg/kg maximum 1.6 mg/dose 4 hour dose limit 0.24-0.3 mg/kg (Maximum dosing will not exceed 25 mg/4 hrs).
  Arms: Randomization to Nubain

SUMMARY:
The pathophysiology of sickle cell disease (SCD) manifestations, are complex with interactions of intracellular hemoglobin, membrane and endothelial activation but the hallmark remains recurrent and painful vaso-occlusive episodes (VOC). These painful episodes are thought to result from ischemia caused when small blood vessels are occluded by misshapen, inflexible erythrocytes. Painful episodes are the most common cause of hospitalization, morbidity, and impairment for SCD patients. There is no therapy that completely prevents or directly aborts painful events for all patients. Consequently, treatment for acute VOC is primarily supportive using hydration and medicinal pain control. Every pain medication has the potential to relieve pain but is associated with significant limitations and side effects.

The primary hypothesis to be tested in this double blind, randomized controlled trial is that Nalbuphine is equivalent to morphine for pain control and patients will suffer fewer episodes of acute chest syndrome. The investigators also expect subjects will report fewer side effects from respiratory depression, abdominal distention from reduced peristalsis, reduced histamine release causing pruritis and still be provided adequate pain control. Further hypotheses to be tested is ability to recruit patient participants while being treated in the Emergency Department and that continuous infusion of Nalbuphine with accompanying patient controlled analgesia (PCA) is safe and effective in controlling pain, requiring less total opiates consumption, while decreasing length of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease (SS, SC, SβThal) who are hospitalized for acute painful episodes
* 6 years old and < 19 years old
* Normal baseline chest radiograph
* Normal renal and hepatic function within the previous 12 months

Exclusion Criteria:

* Previous patient participation in this clinical trial
* Any patient on chronic transfusion Any patient with pulmonary infiltrate on chest radiograph on admission
* Any patient with DSM diagnosis, excluding those with Attention Deficit Disorder, on or off treatment
* Any patient with documented allergy to either study drug
* Any patient with known evidence of an underlying disease that would interfere with evaluation of a therapeutic response such as:

  * Hepatic dysfunction (3x ALT),
  * Renal dysfunction (Cr > 1 children/adolescents, Cr >2 adults),
  * Pulmonary Hypertension (TRJ >3.0),
  * Cardiac dysfunction.
  * Any patient with symptoms of an acute stroke.
  * Any patient known or suspected to be pregnant.
  * Any patient with priapism
  * The patient or guardian who will not give consent or assent to be randomized.

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05-26 (Actual); Primary Completion 2014-01-14 (Actual); Study Completion 2016-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Randomizing Particiipants to Morphine: Randomizing participants to Morphine or Nubain for treatment of Sickle Cell Pain Crisis
  Morphine: Loading Dose: 0.1mg/kg. May repeat every 15 min up to a maximum of 3 total doses until pain controlled.
  Continuous rate: 0.01-0.04mg/kg/hr (titrated to comfort level) PCA dose 0.01-0.03 mg/kg maximum 1.6 mg/dose 4 hour dose limit 0.24-0.3 mg/kg (Maximum dosing will not exceed 25 mg/4 hrs).
- Randomization to Nubain: Randomization toNubain or Morphine for the management of Pain Crisis in Sickle Cell patients
  Nubain: Loading Dose: 0.1mg/kg. May repeat every 15 min up to a maximum of 3 total doses until pain controlled.
  Continuous rate: 0.01-0.04mg/kg/hr (titrated to comfort level) PCA dose 0.01-0.03 mg/kg maximum 1.6 mg/dose 4 hour dose limit 0.24-0.3 mg/kg (Maximum dosing will not exceed 25 mg/4 hrs).
Period: Overall Study
Arm/Group | Randomizing Particiipants to Morphine | Randomization to Nubain
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomizing Particiipants to Morphine | Randomization to Nubain | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 8 | 13 | 21
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Acute Chest Syndrome
Description: Number of Participants with Acute Chest Syndrome or A new pulmonry infiltrate on Chest X-ray
Time Frame: 3 days
Measure: Number; unit: participants
Arm/Group | Randomizing Particiipants to Morphine | Randomization to Nubain
Number analyzed (Participants) | 20 | 20
participants | 2 | 1

2. Secondary Outcome: Number of Participants Who Experienced Pain Relief
Time Frame: 2 days
Measure: Number; unit: participants
Arm/Group | Randomizing Particiipants to Morphine | Randomization to Nubain
Number analyzed (Participants) | 20 | 20
participants | 2 | 2

ADVERSE EVENTS:
Arm/Group | Randomizing Particiipants to Morphine | Randomization to Nubain
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No